CLINICAL TRIAL: NCT01028248
Title: Phase I, Open-Label, Single-Center, Randomized, Study of the Safety and Efficacy of 0.5 mg and 2.0 mg Ranibizumab in Patients With Macular Edema Secondary to Perfused Central Retinal Vein Occlusion
Brief Title: Lucentis for Macular Edema Associated With Central Retinal Vein Occlusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Dante J. Pieramici, California Retina Consultants and Research Foundation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FVF4714s
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Central Retinal Vein Occlusion
Keywords: Central Retinal Vein Occlusion; Retinal Vein Occlusive disease
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2.0 mg Ranibizumab (Active Comparator)
  Interventions: Drug: Ranibizumab (Lucentis)
- 0.5 mg Ranibizumab (Active Comparator)
  Interventions: Drug: Ranibizumab (Lucentis)

INTERVENTIONS:
Drug: Ranibizumab (Lucentis) — 0.5mg and 2.0mg dose of Ranibizumab 0.05ml administered intravitreally

SUMMARY:
The purpose of this study is to determine whether ranibizumab (Lucentis) will be effective in reducing if not eliminating the macular edema associated with the disease, central retinal vein occlusion (CRVO).

DETAILED DESCRIPTION:
Retinal Venous Occlusive disease is the second only to diabetic retinopathy as a major cause of blindness associated with retinal vascular disease. Macular edema is a major cause of vision loss in patients presenting with central and hemi vein occlusions. Until recently the standard of care for macular edema secondary to central retinal vein occlusion was observation. Recent investigations of steroids for this condition has shown greater visual benefit but is associated with risks such as cataract formation and increased intraocular pressure. In the past laser photocoagulation has been used, but was found to offer no visual benefits over the natural history in the treatment of macular edema associated with CRVO.

Ranibizumab (rhuFab V2), an anti-VEGF agent, is a potent inhibitor of vascular permeability, with the potential to reduce retinal vascular leakage and diminish macular edema. In addition, as an anti-VEGF agent, it may also inhibit neovascularization of the iris, a frequent complication of ischemic central retinal vein occlusion. Ranibizumab use as an intravitreal agent does carry the risk of intraocular infection but probably carries very low risk of glaucoma or cataract formation, making it a potentially safer pharmacologic treatment for CRVO associated macular edema as compared to steroids.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Clinical evidence of perfused central retinal vein occlusion. A central retinal vein occlusion (CRVO) is defined as an eye that has retinal hemorrhages and a dilated retinal venous system in all 4 quadrants. Other evidence of a CRVO may include telangiectatic capillary bed and collateral vessels at the optic nerve head.
* Central macular edema present on clinical examination and OCT testing with a central point thickness and/or central 1mm subfield thickness > 250 microns.
* Visual acuity score greater than or equal to 19 letters (20/400) and less than or equal to 73 letters (20/40) by the ETDRS visual acuity protocol.
* Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or known to be pregnant; also pre-menopausal women not using adequate contraception.
* Participation in another ocular investigation or trial simultaneously
* Uncontrolled hypertension
* Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g. chronic alcoholism, drug abuse)
* Significant diabetic retinopathy (greater than moderate NPDR) or macular edema associated with diabetic retinopathy
* Evidence of vitreoretinal interface abnormality after ocular exam or OCT that may be contributing to the macular edema
* An eye that, in the investigator's opinion, has no chance of improving in visual acuity following resolution of macular edema (e.g. presence of subretinal fibrosis or geographic atrophy)
* Presence of another ocular condition that may affect the visual acuity or macular edema during the course of the study (e.g. AMD, uveitis, Irvine-Gas)
* Evidence of neovascularization of the iris or retina (presence of ischemic CRVO)
* Evidence of central atrophy or fibrosis in the study eye
* Presence of substantial cataract, one that might decrease the vision by 3 or more lines of vision at sometime during the study.
* History of grid/focal laser or panretinal laser in the study eye
* History of vitreous surgery in the study eye
* History of use of intravitreal, peribulbar, or retrobulbar steroids within six months of the study.
* History of cataract surgery within 6 months of enrollment.
* History of YAG capsulotomy within 2 months of the surgery.
* Visual acuity <20/400 in the fellow eye
* Uncontrolled glaucoma (pressure >30) despite treatment with glaucoma medications.
* History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be mean change from baseline best-corrected visual acuity, at Months 6 and 12, based on ETDRS visual acuity chart assessment starting distance of 4 meters. | 6 months and 12 months

SECONDARY OUTCOMES:
Mean number of treatments up to and including Month 6 and 12 for each group (0.5-mg and 2.0-mg). | 6 months, 12 months
Mean change from baseline in center point thickness, central 1mm subfield thickness and total macular volume over time as measured as assessed by spectral-domain or fourier-domain OCT up to Month 12. | 12 months
To determine if changes in mean best-corrected visual acuity are correlated with changes in total macular volume, center point thickness, and/or central 1mm subfield thickness. | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dante J Pieramici, MD, Principal Investigator — California Retina Consultants
Locations (3):
- United States (3):
  - California Retina Consultants, Bakersfield, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California